CLINICAL TRIAL: NCT06253182
Title: Psychosexual Educational Partners Program (PEPP): Randomized Phase II Trial
Brief Title: Psychosexual Educational Partners Program (PEPP)
Acronym: PEPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UTK IRB-23-07925-XP
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Gynecologic Cancer; Sexual Dysfunction; Partner Communication
Keywords: breast cancer; gynecologic cancer; sexual dysfunction; partner communication; couples; intimacy; sexual health
MeSH Terms: conditions — Breast Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized controlled trial
Who Masked: Participant
Masking Description: single masking, participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Guided PEPP Intervention workbook (Experimental): Following completion of the virtual consent/baseline visit and the virtual education visit, dyads will work through content of self-guided workbook. Every two weeks, participants will receive a check-in email and/or text message from study staff to assess their adherence and respond to questions or concerns.
  Interventions: Behavioral: Self-Guided PEPP Intervention Workbook
- Self-Guided PEPP Education Workbook (Active Comparator): Following completion of the virtual consent/baseline visit and the virtual education visit, dyads will work through content of self-guided workbook. Every two weeks, participants will receive a check-in email and/or text message from study staff to assess their adherence and respond to questions or concerns.
  Interventions: Behavioral: Self-Guided PEPP Education Workbook

INTERVENTIONS:
Behavioral: Self-Guided PEPP Intervention Workbook — The workbook contains 3 modules. To complete the workbook in six weeks (one module every 2 weeks), it is recommended that a dyad schedule at least three 30-minute blocks of time each week. Dyads are asked to work through the modules in order and encouraged to set a pace that works for them.
  Arms: Self-Guided PEPP Intervention workbook
Behavioral: Self-Guided PEPP Education Workbook — The workbook contains 3 modules. To complete the workbook in six weeks (one module every 2 weeks), it is recommended that a dyad schedule at least three 30-minute blocks of time each week. Dyads are asked to work through the modules in order and encouraged to set a pace that works for them.
  Arms: Self-Guided PEPP Education Workbook

SUMMARY:
The purpose of this study is to compare two Psychosexual Educational programs for women who have completed treatment for breast or gynecological cancer and their partners in preparation for a well-powered phase III study. The investigators plan to enroll 30 dyads in a 2-arm pilot randomized controlled trial (RCT).

The primary aim will be to assess the preliminary efficacy of the Psychosexual Educational Partners Program (PEPP) on sexual communication.

DETAILED DESCRIPTION:
The Psychosexual Educational Partners Program (PEPP) is a two-arm pilot randomized controlled trial that will compare two approaches to a self-paced, workbook-based intervention. PEPP was designed to enhance intimacy among breast and gynecological cancer survivors and their partners by improving sexual communication. The primary aim of the study is to assess the preliminary efficacy of the revised PEPP intervention on sexual communication. Secondary aims include assessing the preliminary efficacy of PEPP on self-efficacy to communicate about sex and intimacy among cancer survivors; and evaluating adherence, acceptance and adverse events within each study arm.

The intervention is six weeks long and does not require any in-person visits. If a breast or gynecological cancer survivor is determined eligible, they will be educated on the purpose, requirements, and procedures. If interested, participants will be emailed the consent form and will schedule a virtual consent/baseline visit that will include their partner. After consent is obtained from both partners, the dyad will be randomly assigned to a study arm and given study numbers. Both members of the dyad will complete online surveys at the virtual baseline visit. The PEPP workbook will be sent to the participants' address and a virtual education visit will be scheduled. At this second virtual visit, both members of the dyad will receive education about their study arm and a start date will be agreed upon for week 1. Beginning week 1 and continuing through week 6, dyads will work through the PEPP workbook which contains three modules. Participants will receive a scheduled email and/or text check-in message from study staff every two weeks to coincide with the end of each module. Messages will provide a link to a brief survey to assess adherence and respond to any participant questions or concerns. Online surveys will be repeated and adverse events will be assessed at week 6.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 female.
2. Able to read and write in English.
3. History of any stage of breast and/or gynecological cancer.
4. Completed primary treatment (chemotherapy, radiation and/or surgery) ≥ 3 months and ≤ 10 years prior to registration.
5. May use maintenance therapy and concurrent adjuvant endocrine therapy or human epidermal growth factor receptor 2 negative (HER2-) targeted therapy while on study.
6. Have a stable partner, defined as anyone with whom the woman has had an intimate relationship for at least 3 months prior to her cancer diagnosis.
7. Responds yes to the question "Has there been a change in communication and/or intimacy with your partner since your cancer diagnosis?"
8. Both partner and woman patient must agree to participate in the study and sign informed consent to the study.
9. Psychiatric medications such as antidepressants and benzodiazepines are allowed if a person has been on them for 30 days prior to registration, and dose or treatment is not expected to change.

Exclusion Criteria:

1. Past history of sexual abuse.
2. Uncontrolled psychiatric disorder such as major depressive disorder, bipolar disorder, obsessive compulsive disorder, or schizophrenia (Defined per medical history and/or patient self-report).
3. Currently enrolled in another study that addresses sexual health (enrollment in other clinical trials will be allowed).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must be female breast or gynecological cancer survivors and their intimate partners.
Enrollment: 60 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dyadic Sexual Communication (DSC) | consent through study completion, an average of 8 weeks
  The preliminary efficacy of the revised PEPP intervention on sexual communication among dyads. The DSC is a single-dimensional 13-item scale that measures sexual communication between partners on a 4-point Likert scale, disagree strongly to agree strongly. Possible scores range from 13-52 with higher scores indicating better sexual communication.

SECONDARY OUTCOMES:
Self-Efficacy to Communicate about Sex and Intimacy (SECSI) | consent through study completion, an average of 8 weeks
  The SECSI is a is a 10-item scale that measures self-efficacy to communicate about sex and intimacy among women treated for cancer. Participants respond using a 4-point Likert scale, strongly agree to strongly disagree. Possible scores range from 0-30 with higher scores indicating greater self-efficacy to communicate with a partner about sex and intimacy after cancer treatment.
Adherence rate | consent of first participant through study completion of last participant, up to 1 year
  The number of PEPP modules completed by participants divided by the number of participants multiplied by 3 (the total number of modules).
Adverse events | consent through study completion, an average of 8 weeks
  Evaluate the adverse events in participants randomized to each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Noel M Arring, DNP, PhD, RN, Principal Investigator — University of Tennessee Knoxville
Locations (1):
- University of Tennessee Knoxville, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study and as such, data will be thoroughly interrogated. However, if an investigator feels there are unanswered questions or wishes to add to a larger dataset, we would entertain all data-sharing requests for de-identified data as appropriate.